CLINICAL TRIAL: NCT02574091
Title: A Single-Center, Randomized, Double-blind, Placebo-Controlled Study to Evaluate Safety, Tolerability and Pharmacokinetics of Icotinib Hydrochloride Cream in Healthy Adult Participants, Followed by Patients With Mild to Moderate Psoriasis
Brief Title: Icotinib Hydrochloride Cream in Healthy Adults and Psoriasis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BD-ICC-NZ-I01
Record Dates: First submitted 2015-09-28; First posted 2015-10-12 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Psoriasis
Keywords: EGFR inhibitor; topical agent; psoriasis; phase 1
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cohort 1-Experimental (Experimental): 4 healthy adult participants will be randomized to receive 1% icotinib hydrochloride cream, applied twice daily for 7 consecutive days (final dose on the morning of Day 8).
  The drug will be used topically to the back of each participant within an area of 15cm x 25cm.
  Interventions: Drug: 1% icotinib hydrochloride cream
- Cohort 1-Placebo (Placebo Comparator): 2 healthy adult participants will be randomized to receive placebo (blank cream), applied twice daily for 7 consecutive days (final dose on the morning of Day 8).
  The drug will be used topically to the back of each participant within an area of 15cm x 25cm.
  Interventions: Drug: Placebo
- Cohort 2-Experimental (Experimental): 4 healthy adult participants will be randomized to receive 2% icotinib hydrochloride cream, applied twice daily for 7 consecutive days (final dose on the morning of Day 8).
  The drug will be used topically to the back of each participant within an area of 15cm x 25cm.
  Interventions: Drug: 2% icotinib hydrochloride cream
- Cohort 2-Placebo (Placebo Comparator): 2 healthy adult participants will be randomized to receive matching placebo, applied twice daily for 7 consecutive days (final dose on the morning of Day 8).
  The drug will be used topically to the back of each participant within an area of 15cm x 25cm.
  Interventions: Drug: Placebo
- Cohort 3-Experimental (Experimental): 6 patients with mild to moderate psoriasis will be randomized to receive 1% icotinib hydrochloride cream, applied twice daily for 13 consecutive days (final dose on the morning of Day 14).
  The drug will be applied topically to the psoriasis site (excluding face, scalp, genital and groin) on the arms and/or legs and/or trunk only.
  Interventions: Drug: 1% icotinib hydrochloride cream
- Cohort 3-Placebo (Placebo Comparator): 2 patients with mild to moderate psoriasis will be randomized to receive matching placebo, applied twice daily for 13 consecutive days (final dose on the morning of Day 14).
  The drug will be applied topically to the psoriasis site (excluding face, scalp, genital and groin) on the arms and/or legs and/or trunk only.
  Interventions: Drug: Placebo
- Cohort 4-Experimental (Experimental): 6 patients with mild to moderate psoriasis will be randomized to receive 2% icotinib hydrochloride cream, applied twice daily for 13 consecutive days (final dose on the morning of Day 14).
  The drug will be applied topically to the psoriasis site (excluding face, scalp, genital and groin) on the arms and/or legs and/or trunk only.
  Interventions: Drug: 2% icotinib hydrochloride cream
- Cohort 4-Placebo (Placebo Comparator): 2 patients with mild to moderate psoriasis will be randomized to receive matching placebo, applied twice daily for 13 consecutive days (final dose on the morning of Day 14).
  The drug will be applied topically to the psoriasis site (excluding face, scalp, genital and groin) on the arms and/or legs and/or trunk only.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1% icotinib hydrochloride cream — Topical administration for twice daily
  Other Names: no other name
  Arms: Cohort 1-Experimental; Cohort 3-Experimental
Drug: 2% icotinib hydrochloride cream — Topical administration for twice daily.
  Other Names: no other name
  Arms: Cohort 2-Experimental; Cohort 4-Experimental
Drug: Placebo — Topical administration for twice daily.
  Other Names: Blank Cream
  Arms: Cohort 1-Placebo; Cohort 2-Placebo; Cohort 3-Placebo; Cohort 4-Placebo

SUMMARY:
This is a phase I study to evaluate the safety, tolerability and pharmacokinetics of Icotinib Hydrochloride Cream in healthy adults and patients with mild to moderate psoriasis.

DETAILED DESCRIPTION:
Icotinib Hydrochloride is a small-molecule epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor, which has been approved for the treatment of advanced non-small-cell lung cancer (NSCLC) in China in its oral form. As EGFR is implicated in the pathogenesis of psoriasis, icotinib hydrochloride is being developed as a cream for the treatment of mild to moderate psoriasis. This is a single-center, randomized, double-blind, placebo-controlled study of icotinib hydrochloride cream by topical administration. The study is designed in two parts in healthy subjects (part 1) followed by patients with mild to moderate psoriasis (part 2). 1% and 2% icotinib hydrochloride cream will be initially applied to healthy subjects. Once the study in healthy adults shows favorable safety and tolerability, a study in patients with mild to moderate psoriasis will be followed. Approximately 28 subjects will be enrolled, including 12 healthy subjects (Part 1) and 16 patients with psoriasis (Part 2).

ELIGIBILITY:
Inclusion Criteria:

For Part 1-Healthy Participants

* 18-50 years old (inclusive), male or female
* Male participants should be ≥ 50 kg, female participants should be ≥ 45 kg; Body Mass Index (BMI) should be between 19 and 30 kg/m2 (inclusive)
* In good health, with no history of diseases of major organs and no BP, HR, ECG or respiratory abnormality on physical examination
* Adequate hepatic and renal function, as determined by clinical laboratory assessments of blood and urine
* Negative serum pregnancy test at Screening and negative urine pregnancy test at Day -1 for females of child bearing potential
* Negative screen for drugs of abuse, alcohol, hepatitis B surface antigen (HBsAg), hepatitis C (HCV) and Human Immunodeficiency Virus (HIV) at screening; and negative drugs of abuse, alcohol pre dose on Day -1
* Have signed a written informed consent before entering the study

For Part 2 - Patients with Psoriasis

* Clinical diagnosis of psoriasis for at least six months with multiple affected areas (excluding the face, scalp, genitals and groin) involving 2%-15% of the total Body Surface Area (BSA)
* 18-65 years old
* Male participants should be ≥ 50 kg, female participants should be ≥ 45 kg; BMI should be between 19 and 35 kg/m2 (inclusive)
* In good health, with no history of diseases of major organs and no BP, HR, ECG or respiratory abnormality on physical examination
* Adequate hepatic and renal function, as determined by clinical laboratory assessments of blood and urine
* Negative serum pregnancy test at Screening and negative urine pregnancy test at Day -1 for females of child bearing potential
* Negative screen for drugs of abuse, alcohol, HBsAg, HCV and HIV at screening; and negative drugs of abuse, alcohol pre dose on Day1
* Women of child-bearing potential must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 90 days following completion of therapy
* Have signed a written informed consent before entering the study

Exclusion Criteria:

For Part 1-Healthy Participants

* Any clinically significant central nervous system, cardiac, pulmonary, renal, gastrointestinal, respiratory, metabolic conditions (or history), or other pathological or physiological conditions that might interfere with the trial result
* History of postural hypotension
* Use of any topical agents (including non-medicated lotions such as sun screen, cosmetics, moisturizing lotion) at the administration site within a week before randomization
* History of serious skin diseases (as determined by the investigator); no presence of skin ulceration at the test area at the time of the Screening visit
* Current smoker, or a history of regular (more than weekly) use of tobacco- or nicotine-containing products within two months prior to screening
* History of excessive alcohol intake (more than four standard drinks daily, on average) or use of recreational drugs within the last three months

For Part 2 - Patients with Psoriasis

* Any clinically significant central nervous system, cardiac, pulmonary, renal, gastrointestinal, respiratory, metabolic conditions (or history), or other pathological or physiological conditions that might interfere with the trial result
* History of postural hypotension
* Use of any topical agents (including non-medicated lotions such as sun screen, cosmetics, moisturizing lotion) at the administration site within a week before randomization
* History of serious skin diseases (as determined by the investigator); no presence of skin ulceration at the test area at the time of the Screening visit
* Excessive smoker(≥10 cigarettes per day), or a history of regular (more than weekly) use of tobacco- or nicotine-containing products within two months prior to screening
* History of excessive alcohol intake (more than four standard drinks daily, on average) or use of recreational drugs within the last three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-11-26 (Actual); Primary Completion 2017-02-19 (Actual); Study Completion 2017-02-19 (Actual)

PRIMARY OUTCOMES:
Adverse events in healthy subjects | 8 days
  Incidence and severity of Adverse Events (AE) Vital signs (temperature, Heart Rate (HR), BP and respiration); Clinical laboratory assessments (serum chemistry, hematology and urinalysis); ECG; Use of concomitant medications
Adverse events in patients with mild to moderate psoriasis | 14 days
  Incidence and severity of AEs; Vital signs (temperature, HR, BP and respiration); Clinical laboratory assessments (serum chemistry, hematology and urinalysis); ECG; Use of concomitant medications

SECONDARY OUTCOMES:
Tolerance-related skin reactions in healthy adult participants at the tested sites | 8 days
  Skin irritation and allergy observation (including redness, swelling, itching, pain)
Tolerance-related skin reactions in patients with mild to moderate psoriasis at the tested sites | 14 days
  Skin irritation and allergy observation (including redness, swelling, itching, pain)
To investigate peak plasma concentration (Cmax) of single-dose Icotinib Hydrochloride Cream in healthy adult participants | 8 days
To investigate time maximum concentration observed(tmax) of single-dose Icotinib Hydrochloride Cream in healthy adult participants | 8 days
To investigate area under the plasma concentration versus time curve(AUC) of single-dose Icotinib Hydrochloride Cream in healthy adult participants | 8 days
  AUClast, AUC0-inf will be assessed
To investigate half life(t1/2) of single-dose Icotinib Hydrochloride Cream in healthy adult participants | 8 days
To investigate stable peak plasma concentration (Cmaxss) of repeat-dose Icotinib Hydrochloride Cream in healthy adult participants | 8 days
To investigate time maximum concentration observed(tmax) of repeat-dose Icotinib Hydrochloride Cream in healthy adult participants | 8 days
To investigate area under the plasma concentration versus time curve(AUC) of repeat-dose Icotinib Hydrochloride Cream in healthy adult participants | 8 days
  AUC0-12,AUClast, AUC0-inf will be assessed
To investigate half life(t1/2) of repeat-dose Icotinib Hydrochloride Cream in healthy adult participants | 8 days
To investigate peak plasma concentration (Cmax) of single-dose Icotinib Hydrochloride Cream in patients with mild to moderate psoriasis | 14 days
To investigate time maximum concentration observed(tmax) of single-dose Icotinib Hydrochloride Cream in patients with mild to moderate psoriasis | 14 days
To investigate area under the plasma concentration versus time curve(AUC) of single-dose Icotinib Hydrochloride Cream in patients with mild to moderate psoriasis | 14 days
  AUClast, AUC0-inf will be assessed
To investigate half life(t1/2) of single-dose Icotinib Hydrochloride Cream in patients with mild to moderate psoriasis | 14 days
To investigate stable peak plasma concentration (Cmaxss) of repeat-dose Icotinib Hydrochloride Cream in patients with mild to moderate psoriasis | 14 days
To investigate time maximum concentration observed(tmax) of repeat-dose Icotinib Hydrochloride Cream in patients with mild to moderate psoriasis | 14 days
To investigate area under the plasma concentration versus time curve(AUC) of repeat-dose Icotinib Hydrochloride Cream in patients with mild to moderate psoriasis | 14 days
  AUC0-12,AUClast, AUC0-inf will be assessed
To investigate half life(t1/2) of repeat-dose Icotinib Hydrochloride Cream in healthy adult participants | 14 days
Psoriasis Area and Severity Index (PASI) Scores in patients with mild to moderate psoriasis | 14 days
Dose-toxicity correlation in single-dose and repeat-dose administration | 14 days
  If observable trends exist between dose applied (in Part 2 of the study) and toxicity and response parameters.
Dermatology Life Quality Index (DLQI) | 14 days
Dose-response correlation in single-dose and repeat-dose administration | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Wynne, Study Chair — Christchurch Clinical Studies Trust
Locations (1):
- Christchurch Clinical Studies Trust, Christchurch, New Zealand